CLINICAL TRIAL: NCT02778568
Title: Acute Cardiovascular Responses and Chronic Adaptations of Strength Exercise in Intermittent Claudication Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Raphael M. Ritti Dias, Full Professor, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMR2013FCPE MOVED
Record Dates: First submitted 2013-12-12; First posted 2016-05-20 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Resistance Training; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Training (Experimental): Patients performed resistance exercises
  Interventions: Behavioral: Resistance training
- Control (Active Comparator): Patients who performed flexibility exercise
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Resistance training — Resistance training exercises
  Other Names: Physical training
  Arms: Resistance Training
Behavioral: Control — Stretching exercises
  Arms: Control

SUMMARY:
The aim of this study was to analyze the effects of resistance exercise and training on cardiovascular function of peripheral artery disease patients.

DETAILED DESCRIPTION:
Several studies have shown that strength training can promote important benefits for the cardiovascular system in healthy subjects and patients with chronic diseases. However, the effects of resistance exercise on cardiovascular function in intermittent claudication patients are unclear. In addition, it also do not know the chronic effects on cardiovascular function in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Had a graded treadmill test that was limited by claudication (2 minutes)
* Had an ankle brachial index <0.90
* Had systolic blood pressure ,160 mmHg and/or diastolic blood pressure,105 mmHg
* Were not performing any regular exercise program
* Were not using antihypertensive medications affecting the heart rate (e.g., b-blockers and nondihydropyridine calcium channel blockers)
* Were nonobese
* Individuals who have not undergone bypass surgery or angioplasty least one year ago

Exclusion Criteria:

* Had no symptoms related to myocardial ischemia during the treadmill test
* Amputation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Change from baseline to 12 and 24 weeks

SECONDARY OUTCOMES:
Change in Walking distance | Change from baseline to 12 and 24 weeks
Change in Health related Quality of life | Change from baseline to 12 and 24 weeksBaseline, 12 wks and 24 wks
Change in Muscle blood flow of limbs | Change from baseline to 12 and 24 weeks
  Muscle blood flow assessed with venous occlusion plethysmography
Change in body fat | Change from baseline to 12 and 24 weeks
Change Serum Cholesterol | Change from baseline to 12 and 24 weeks
Change in serum glucose | Change from baseline to 12 and 24 weeks
Change in TNFalpha | Change from baseline to 12 and 24 weeks
Change in Score Short-physical performance battery | Change from baseline to 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marilia A Correia, MS, Study Chair — University of Pernambuco
Locations (1):
- Emergency Hospital of Pernambuco - PROCAPE, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No